CLINICAL TRIAL: NCT01803308
Title: A Phase 1a/1b Multiple Ascending Dose Study to Assess the Safety, Pharmacokinetics and Pharmacodynamics of SB 9200 in Treatment Naïve HCV Infected Adults
Brief Title: A Multiple Ascending Dose Phase I Study of SB 9200 in Treatment Naïve Adults With Chronic Hepatitis C Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syneos Health (Other)
Collaborators: F-star Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SB12-9200-101
Record Dates: First submitted 2013-02-27; First posted 2013-03-04 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2014-08

CONDITIONS: Hepatitis C Infection
Keywords: Hepatitis C Infection; Treatment Naïve, Chronic; First In Human; Single Ascending Dose; Multiple Ascending Dose
MeSH Terms: conditions — Hepatitis C; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Part A (Experimental): Experimental: Part A: Part A will use a single ascending dose protocol in small, open-label cohorts to determine the starting dose for Part B in the potentially therapeutic range.
  Intervention: SB9200
  Interventions: Drug: SB9200
- Experimental Part B (Experimental): Experimental: Part B: Part B will use a multiple ascending dose protocol to further explore the safety, tolerability, pharmacokinetics and pharmacodynamics of SB9200 over 7-14 days of dosing.
  Intervention: SB9200 and Placebo
  Interventions: Drug: SB9200; Drug: Placebo

INTERVENTIONS:
Drug: SB9200 — Part A open-label, single ascending doses of SB9200 from 100mg - 1500mg.
  Arms: Experimental Part A
Drug: SB9200 — Part B randomised 6:2 (active:placebo) using recommended Part B starting dose, and ascending to up to 1500mg for 7-14 days of dosing.
  Arms: Experimental Part B
Drug: Placebo — Part B randomised 6:2 (active:placebo) using anhydrous lactose capsules identical to active comparator, minus active ingredient.
  Arms: Experimental Part B

SUMMARY:
The purpose of this study is to compare the safety and tolerability of ascending doses of SB 9200 given for up to 14 days to subjects with chronic Hepatitis C infection.

DETAILED DESCRIPTION:
This is a First-in-human, Two-stage, Multi-centre study. Part A is an open-label, single ascending dose study in fed or fasted subjects and Part B is a randomized, placebo-controlled multiple ascending dose study. The study is designed to evaluate the safety and tolerability of ascending doses of SB 9200 given as monotherapy for up to 14 days to subjects with chronic Hepatitis C infection, and to determine the pharmacokinetic and pharmacodynamic relationship over this dose range.

ELIGIBILITY:
Inclusion Criteria:

* Must provide written informed consent before any assessment is performed.
* Must be willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Males or females of non-childbearing potential between the ages of 18 and 60 years, inclusive.
* Must have HCV and laboratory evidence of HCV infection for at least six months before the Screening Visit.
* Must have HCV-1 (1a or 1b or non-sub-typeable HCV-1), HCV-2 or HCV-3, as applicable for a given cohort.
* Subjects must have a plasma HCV RNA >5 log10 IU/mL (100,000 IU/mL).
* Must have fibrosis of Stage 2 or lower by Ishak or Metavir scoring system or equivalent as evidenced by a recent (within two years of screening) liver biopsy (i.e. no more than moderate fibrosis). If a recent liver biopsy is not available, Fibroscan of < 8.5 kilopascals at screening.
* Must have negative human immunodeficiency virus (HIV) and Hepatitis B screening test results.
* Must have a body mass index (BMI) of 18-32 kg/m2 (inclusive).
* Must have screening laboratory values within the reference ranges or if outside the normal range, not clinically significant as judged by the Investigator. ALT and aspartate aminotransferase (AST) must be within 2x the upper limit of normal.
* Must not consume grapefruit or grapefruit-related citrus fruits or juice from seven days prior to the first dose of study drug until collection of the final PK blood sample at 14 days after the last dose of study drug.
* Must be able to communicate with site personnel and understand instructions.

Exclusion Criteria:

* Any previous treatment with an investigational or approved drug or drug regimen for the treatment of HCV. Note: SB 9200 is excluded from this criterion, i.e. subjects who complete Part A of the study will be eligible to participate in Part B of the study.
* History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes.
* Use of nonprescription drugs, vitamins and dietary supplements within 14 days or five half-lives (whichever is longer) prior to the trial dose medication. Changes to prescription medication within 14 days prior to the first dose of study medication (i.e. only stable prescription medications are permitted whilst on study).
* History of intercurrent illness (e.g., upper respiratory illness with fever) within five days prior to the first dose of study drug.
* History of illicit or controlled substance abuse or alcohol abuse within one year before the Screening Visit (with the exception of cannabinoids).
* Any condition possibly affecting drug absorption (e.g., gastrectomy).
* Long QT syndrome or QTc > 450 msec for males and > 470 msec for females at screening or baseline.
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past five years, regardless of whether there is evidence of local recurrence or metastases.
* Women of child-bearing potential.
* Fertile males, defined as all males physiologically capable of conceiving offspring unless the subject and partner of child bearing potential agree to comply with acceptable contraception and the female partner is not lactating.
* Prior liver biopsy (at any time in the past), indicating Stage 3 or higher fibrosis by Ishak or Metavir scoring system or equivalent (i.e. greater than moderate fibrosis).
* Any other cause of significant liver disease in addition to HCV, which may include, but is not limited to, malignancy with hepatic involvement, hepatitis B, drug or alcohol related cirrhosis, autoimmune hepatitis, hemochromatosis, Wilson's disease, or primary biliary cirrhosis.
* Evidence or history or clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Blood donation of approximately 500 mL or significant blood loss within 56 days prior to dosing.
* Any other medical or psychiatric condition or laboratory abnormality which, in the view of the Investigator, is likely to interfere with the study or put the subject at risk.
* Concurrent participation in another clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2013-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Safety | Up to 35 days
  Clinical safety data from 12-lead ECG, clinical laboratory tests, urinalysis, treatment-emergent adverse events, vital signs (blood pressure, heart rate, respiratory rate).

SECONDARY OUTCOMES:
Pharmacokinetic profile of SB9200 | Up to 35 days
  Pharmacokinetic parameters and the PK profile of SB 9200 at doses from 100 mg to 1500 mg given for up to 14 days to subjects with Hepatitis C.
Pharmacokinetic and Pharmacodynamic relationship of SB9200 | Up to 35 days
  Correlation between SB9200 exposure and Hepatitis C RNA level at doses from 100 mg to 1500 mg.
Effect of food on exposure of SB 9200 | Up to 35 days
  Comparison of exposure to SB9200 in fed and fasted states.
Short Term Antiviral Efficacy | Up to 35 days
  Short term antiviral efficacy of ascending doses of SB 9200 monotherapy given for up to 14 days to treatment naïve subjects with Hepatitis C.
Viral Resistance | Up to 35 days
  Viral resistance and describe any resistant mutants that appear during Investigational Product administration.
IL28B Genotype | Up to 35 days
  Association of IL28B genotype (CC, CT or TT) with virologic response to SB 9200 at the chosen dose.

OTHER OUTCOMES:
Exploratory: IFN Expression and IFN pathways | Up to 35 days
  Blood samples will be collected for potential exploratory evaluation of correlations between SB9200 dose and Interferon (IFN) expression, and induction of signalling proteins in IFN pathways such as Interferon Regulatory Factor (IRF)-3, IRF-7, Interferon Stimulated Gene 15 (ISG15) and Extra Erythrocytically expressed haemoglobin (EEEH) levels in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Mitchell, Study Director — F-star Therapeutics, Inc.; Alexander Thompson, MD, PhD, Principal Investigator — Nucleus Network, The Alfred Hospital
Locations (4):
- Australia (3):
  - Nucleus Network, Austin Hospital, Heidelberg, Victoria
  - Nucleus Network, The Alfred Hospital, Melbourne, Victoria
  - Linear Clinical Research, The Queen Elizabeth II Medical Centre, Nedlands, Western Australia
- Primorus Clinical Trials Ltd, Christchurch, New Zealand